CLINICAL TRIAL: NCT04736771
Title: A Retrospective Real-world Evidence Study Assessing the Safety and Effectiveness of the Nobel Biocare N1 Concept System.
Brief Title: Study Assessing the Safety and Effectiveness of the Nobel Biocare N1 Concept System.
Acronym: Evolution
Status: Completed | Type: Observational
Sponsor: Nobel Biocare (Industry)
Responsible Party: Sponsor
Other Study IDs: T-193
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Dental Implant
Keywords: implant site preparation tools, implant system

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Standard medical and dental forms from all subjects (i.e., adults ≥18 years old in need of a dental implant) who have been treated for CS Tiger Ultra Implant TCC RP dental implant treatment at the participating Clinics will be reviewed and clinical data will be obtained, only upon the receipt of Ethical Committee's approval and upon subject's signature of the corresponding Informed Consent Form.

All raw study data will be de-identified and corresponding subject information recorded in the data accrual system (e-CRF Smart Trial). Information recorded by the researcher shall not identify the subject and no individually identifiable data elements shall be recorded. The researcher shall receive a link to log in to e CRF system. The researcher will be asked to create an account and every log-in attempt into the system shall be controlled by an unique code. Radiographic measurements of marginal bone level mesial and distal to the implant (at time of surgery, implant loading and 12-months follow-up post-loading) carried out according to the standard practice of the clinic will be collected for the assessment of the marginal bone levels changes. Data will be anonymized before the x-ray collection.

An independent radiologist shall be responsible for the evaluation of the radiographic data. The Sponsor shall send to the radiologist all corresponding radiographic files entitled by study code, clinic and patient number, implant position and implant characteristics (diameter and/or length - where available) together with an Excel sheet where the Radiologist can accurately track the corresponding bone level measurements.

DETAILED DESCRIPTION:
This study is a retrospective observational multi-center study. It will include data from 70 up to 100 subjects, treated with the N1 Concept System. The study will be conducted in up to six European centers (Appendix I - Participating Institutions).

The study will collect clinical and radiographic data related to the surgery and up to 12-months after loading (a time window of ± 3-months is accepted).

Study subjects will be consecutively included provided they meet all of the inclusion criteria and none of the exclusion criteria.

All participating subjects must have signed the Informed Consent Form together with a separate Consent Form regarding personal data processing (if not waived by the corresponding Ethical Committee). Retrospective data collection will only start after signatures have been provided.

The investigator will check subjects' medical and dental chart and assign a study ID number to each subject. The corresponding study required information will be de-identified and entered into the electronic study database.

All x-ray images, from the area of treatment, that were made up until 12-months after implant loading will be de-identified before uploaded to the study database or otherwise sent to the sponsor.

No personal/confidential information (e.g.: full name or initials, date of birth, social security number, etc.) that could reveal subject's identity will be recorded in the study database.

Endpoints

Primary endpoint The primary endpoint is to evaluate the marginal bone level change of the N1 Concept System from loading to 12-months post loading. Patients with matched readable radiographs are included.

Secondary endpoints

* Implant survival and success rates at 12-months after loading.
* Soft tissue healing parameters (i.e. bleeding index, plaque index, etc.) at 12-months after loading.
* Safety recorded by AE, SAE, ADE, SADE, USADE, and DD.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥18 years of age
* Signed of Informed Consent Form*
* Signed Personal Data Processing (GDPR) Form**
* Subject received Nobel Biocare N1 Concept System implants.

Exclusion criteria: none

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All subjects (i.e., adults ≥18 years old in need of a dental implant) who have been treated for CS Tiger Ultra Implant TCC RP dental implant treatment at the participating Clinics in the period from April 2019 until December 2019 at the corresponding participant Clinics
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-16 (Actual)

PRIMARY OUTCOMES:
Marginal Bone Level and marginal bone levels changes | 12-months post loading

CONTACTS AND LOCATIONS:
Locations (3):
- Urban Dental Center Kft, Budapest, Hungary
- Studio Ban Mancini Fabbri, Cattolica, Italy
- Staas & Bergmans, 's-Hertogenbosch, Netherlands

REFERENCES:
- [Derived] Fabbri G, Staas T, Urban I. A Retrospective Observational Study Assessing the Clinical Outcomes of a Novel Implant System with Low-Speed Site Preparation Protocol and Tri-Oval Implant Geometry. J Clin Med. 2022 Aug 18;11(16):4859. doi: 10.3390/jcm11164859. PMID 36013098